CLINICAL TRIAL: NCT01859767
Title: An Exploratory, Open-label, Non-randomized Phase 1 Study to Evaluate the Efficacy and Safety of MNI-672 SPECT for Detection/Exclusion of Cerebral B-amyloid in Patients With Alzheimer's Disease Compared to Healthy Volunteers.
Brief Title: Efficacy and Safety of MNI-672 SPECT for Detection/Exclusion of Cerebral B-amyloid in AD Subjects Compared to HVs.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Danna Jennings, Principal Investigator, Molecular NeuroImaging
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MNI-672-01
Record Dates: First submitted 2013-04-30; First posted 2013-05-22 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; SPECT
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]MNI-672 SPECT (Experimental): [123I]MNI-672 single photon emission tomography (SPECT)imaging
  Interventions: Drug: [123I]MNI-672 SPECT

INTERVENTIONS:
Drug: [123I]MNI-672 SPECT — Subjects will be dosed by intravenous injection to a target dose of 5 mCi and not to exceed 5.5 (not >10% of 5 mCi limit) I-123 MNI-672 prior to the SPECT scan.
  Other Names: MNI-672

SUMMARY:
This is a Phase 1, single center, open-label, non-randomized, clinical study in probable AD patients and HVs to evaluate the efficacy, safety and tolerability of a single dose of MNI-672. The underlying goal of this study is to assess MNI-672 SPECT imaging as a tool to detect ß amyloid deposition in the brain of AD research participants and young healthy male subjects. All study procedures will be conducted at Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 3 patients with AD and 3 young male HVs will be recruited to participate in this study. HVs will be screened to ensure that there is no evidence of cognitive decline or significant neurological deficit.

All eligible subjects will be required to visit the study center on at least 2 occasions:

1. for one or more screening visits which should include a history and physical examination, laboratory and extensive neuro-psychological testing and MRI brain scanning. AD subjects will also undergo Amyvid PET imaging as part of the Screening Visit.
2. on one day for baseline examinations and MNI-672 administration and subsequent SPECT scanning- followed by safety measures

DETAILED DESCRIPTION:
To determine diagnostic efficacy of the MNI-672 SPECT scans in differentiating between patients with probable AD and HVs on the basis of neocortical tracer binding pattern, the SPECT scans will be visually assessed by a nuclear physician experienced in the field of neuro-imaging. SPECT scan findings will be classified either as abnormal (i.e., significant neocortical uptake in predefined regions) or as normal (i.e. no significant neocortical uptake in predefined regions). The visual analysis of the MNI SPECT images will be compared to the clinical diagnosis and Amyvid PET imaging results to determine the efficacy of MNI-672 as an agent to detect B-amyloid. The nuclear physician evaluating the SPECT images will be unaware of the clinical diagnosis.

ELIGIBILITY:
Healthy Volunteer Inclusion Criteria:

* is male and is 20-30 years of age (inclusive)
* has no evidence of cognitive impairment as indicated by a clinical dementia rating (CDR, [Hughes et al. 1993]) score of 0 (zero) and a score of ≥ 28 in the Mini-Mental Status Examination (MMSE, [Folstein et al. 1975])
* has MRI brain scan that has been judged as "normal (age- appropriate)" including ARWMC scale [Wahlund et al. 2001] scores supporting the lack of cerebrovascular disease (e.g., a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1)
* has no family history of AD defined by more than 1 first-degree relative

Alzheimer disease subject inclusion criteria:

* is male or female and is ≥ 50 of age, whereby females must be without childbearing potential (confirmed by either: age ≥ 60; or history of surgical sterilization or of hysterectomy, or last spontaneous bleeding at least 2 years prior to the study start)
* presents with positive assessment for dementia of Alzheimer's type in accordance with the DSM-IV-TR and probable AD according to the NINCDS-ADRDA criteria and fulfils none of the exclusion criteria of either
* does not fulfill the ICC criteria for probable DLB, the NINDS-AIREN for probable Vascular dementia, or the Neary [Neary et al. 1998] criteria for FTD
* has a CDR [Hughes et al. 1993] score of 0.5, 1 or 2
* MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease (e.g., the ARWMC scale) changes limited to: a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1)
* has an Amyvid PET scan with moderate to frequent amyloid neuritic plaques based on visual interpretation
* has a caregiver who is willing and able to attend study visits and perform the psychometric tests requiring the presence of a caregiver

Exclusion Criteria for all subjects:

* has any contraindication to MRI examination, e.g. metal implants or phobia
* is scheduled for surgery and/or another invasive procedure within the time period of up to 7 days following MNI-672 application
* is medically unstable and whose clinical course during the observation period is unpredictable, e.g. patients / volunteers within 14 days of myocardial infarction or stroke, unstable patients / volunteers with previous surgery (within 7 days), patients with advanced heart insufficiency (NYHA stage IV), or with acute renal failure
* has a history of exposure to any radiation >15 mSv/year (e.g. occupational or radiation therapy)
* is receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)
* has received anti-amyloid drug therapy
* has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening, and/or any radiopharmaceutical within 10 radioactive half-lives prior to MNI-672 administration
* has a brain tumor or other intracranial lesion, a disturbance of CSF circulation (e.g., normal pressure hydrocephalus) and/or a history of serious head trauma or brain surgery
* has a history, physical, laboratory or imaging findings indicative of a significant neurological or psychiatric illness (for patients - other than AD)
* has another disease that can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function)
* has a history of alcohol or drug abuse

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 2 years
  Safety will be assessed by the number of participants with adverse events.
Clinically significant changes in vital signs | 2 years
  Safety will also be assessed by any clinically significant changes in vital signs, ECG parameters, physical examination findings, clinical laboratory findings, and injection site monitoring.

SECONDARY OUTCOMES:
Total I-123 radioactivity in plasma | 2 years
  The plasma concentrations will be expressed in %ID/mL. The I-123 radioactivity will be derived from the concentration -time profile.
Standard uptake values (SUV) | 2 years
  Standard uptake values (SUV) for the target areas including the frontal cortex, temporal cortex, parietal cortex, posterior cingulate cortex and anterior cingulate cortex, and the cerebellum as the reference region will be calculated. Standard uptake values regional (SUVR) for cortical target areas relative to cerebellum will also be calculated.
Visual analysis | 2 years
  The imaging diagnosis will be compared to the clinical diagnosis and Amyvid PET interpretation to determine the efficacy of MNI-672 as a diagnostic tool for AD.

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Molecular NeuroImaging, LLC
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neary D, Snowden JS, Gustafson L, Passant U, Stuss D, Black S, Freedman M, Kertesz A, Robert PH, Albert M, Boone K, Miller BL, Cummings J, Benson DF. Frontotemporal lobar degeneration: a consensus on clinical diagnostic criteria. Neurology. 1998 Dec;51(6):1546-54. doi: 10.1212/wnl.51.6.1546. PMID 9855500
- [Background] Hughes CP et al: A new clinical scale for staging of dementia. British Journal of Psychiatry 1982; 140: 566-572. Updated by Morris J: The CDR: current version and scoring rules. Neurology 1993; 43: 2412-2413
- [Background] Wahlund LO, Barkhof F, Fazekas F, Bronge L, Augustin M, Sjogren M, Wallin A, Ader H, Leys D, Pantoni L, Pasquier F, Erkinjuntti T, Scheltens P; European Task Force on Age-Related White Matter Changes. A new rating scale for age-related white matter changes applicable to MRI and CT. Stroke. 2001 Jun;32(6):1318-22. doi: 10.1161/01.str.32.6.1318. PMID 11387493
- See also: Molecular NeuroImaging, LLC — http://www.mnimaging.com